CLINICAL TRIAL: NCT02129465
Title: Correlates of Maternal Characteristics in CMV Infection in Pregnancy With Maternal-fetal Transmission.
Brief Title: Immunological Characteristics of Maternal-fetal Transmission of Cytomegalovirus in Pregnancy
Acronym: CMV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Yechiel Schlesinger, Head, division of pediatrics, Shaare Zedek Medical Center
Other Study IDs: CMV_transmission.CTIL
Record Dates: First submitted 2014-04-27; First posted 2014-05-02 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Pregnancy; Cytomegalovirus Infections; Congenital Infection
Keywords: Cytomegalovirus; CMV; pregnancy; transmission
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, peripheral blood mono-nuclear cells , DNA, RNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Analysis of several characteristics of blood from pregnant women with CMV infection according to maternal-fetal transmission. These include CMV viral load, cytokine profile in response to in-vitro stimulation with CMV peptides, meticulous analysis of anti CMV antibodies, maternal DNA polymorphism and microarray of gene expression.

DETAILED DESCRIPTION:
Maternal Cytomegalovirus infection in pregnancy may cause significant morbidity in the fetus. Intrauterine CMV transmission occurs mainly during primary maternal infections, with a maternal-fetal transmission rate of about 40%. The mechanisms dictating CMV intrauterine transmission are unknown, and transmission is currently thought to be dependent on multiple factors, including the maternal and fetal immune system.

To investigate the mechanism of transmission approaching laboratory prediction of transmission, the investigators collect blood from pregnant women with primary CMV infection, and analyze several characteristics. These include CMV viral load, cytokine profile in response to in-vitro stimulation with CMV peptides, meticulous analysis of anti CMV antibodies, maternal DNA polymorphism and microarray of gene expression.

These results will be analysed according to transmission as indicated by a positive culture / Polymerase chain transcription of amniotic fluid or newborns urine / saliva.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* CMV infection: primary infection: (1) CMV-specific IgG seroconversion or (2) demonstration of low avidity CMV-specific IgG antibodies, (3) the primary appearance of CMV-specific IgM with no previous IgG, and (4) CMV DNA or viral products in blood Secondary infection: appearance of CMV-specific IgM with positive IgG

Exclusion Criteria:

* CMV status unclear
* spontaneous or induced abortion
* unknown fetal outcome

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with CMV infection who are referred to the 'CMV in Pregnancy clinic' in Shaare Zedek Medical Center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Maternal-fetal transmission of CMV | up to 2 years
  Positive CMV culture and / or PCR in amniotic fluid or newborns urine.

SECONDARY OUTCOMES:
Symptomatic congenital CMV | up to 2 years
  Any clinical findings defining the patient as having symptomatic infection such as microcephaly, intra-cranial calcifications, sensory-neuronal hearing loss, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Schlesinger, MD, Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel; Yifat Eldar-Yedidia, Ph.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel